CLINICAL TRIAL: NCT03422731
Title: Multi-Modality Imaging and Correlative Studies in Patients With Leukemia
Brief Title: Multi-modality Imaging and Collection of Biospecimen Samples in Understanding Bone Marrow Changes in Patients With Acute Myeloid Leukemia Undergoing TBI and Chemotherapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17222; NCI-2017-01778 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17222 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2018-02-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (TMLI+FLT/TMLI) (Experimental): Patients may undergo optional fluorothymidine F-18 PET scan over 2 hours at baseline, on days 30 and 100, at 1 year, and at time of relapse. Patients undergo DECT and water-fat MRI scan over 30 minutes at baseline, on days 30 and 100, at year 1, and at time of relapse. Patients also undergo collection of bone marrow and blood samples at baseline, on days 30 and 100, and at 1 year. Patients undergo fluorothymidine F-18 PET, DECT, and water-fat MRI as in TMLI+FLT.
  Interventions: Procedure: Biospecimen Collection; Procedure: Dual-Energy Computed Tomography; Drug: Fluorothymidine F-18; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Cohort II (TBI) (Active Comparator): Patients undergo collection of bone marrow at baseline, day 30, time of relapse, and at 1 year.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of bone marrow and blood samples
Procedure: Dual-Energy Computed Tomography — Undergo DECT
  Other Names: DECT
  Arms: Cohort I (TMLI+FLT/TMLI)
Drug: Fluorothymidine F-18 — Undergo FLT PET
  Other Names: 18F-FLT; 3''-Deoxy-3''-(18F) Fluorothymidine; 3''-deoxy-3''-[18F]fluorothymidine; ALOVUDINE F-18; Fluorothymidine F 18
  Arms: Cohort I (TMLI+FLT/TMLI)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo water-fat MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
  Arms: Cohort I (TMLI+FLT/TMLI)
Procedure: Positron Emission Tomography — Undergo FLT PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
  Arms: Cohort I (TMLI+FLT/TMLI)

SUMMARY:
This clinical trial investigates multi-modality imaging and collection of biospecimen samples in understanding bone marrow changes in patients with acute myeloid leukemia undergoing total body irradiation (TBI) and chemotherapy. Using multi-modality imaging and collecting biospecimen samples may help doctors know more about how TBI and chemotherapy can change the bone marrow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Temporal assessment of treatment impact on bone marrow. II. Relative assessment of bone marrow status between total marrow and lymphoid irradiation (TMLI) and conventional TBI.

SECONDARY OBJECTIVES:

I. Correlation of dual energy computed tomography (DECT), magnetic resonance imaging (MRI) imaging with biological samples for cellularity/adiposity.

II. Feasibility of fluorothymidine F-18 (FLT) positron emission tomography (PET) imaging biomarker as a predictor of treatment response.

III. Correlation of FLT PET imaging with biological correlate for leukemia. IV. Characterize relative distribution of leukemia in bone marrow (BM) environment.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I (TLMI+FLT/TMLI): Patients may undergo optional fluorothymidine F-18 PET scan over 2 hours at baseline, on days 30 and 100, at 1 year, and at time of relapse. Patients undergo DECT and water-fat MRI scan over 30 minutes at baseline, on days 30 and 100, at year 1, and at time of relapse. Patients also undergo collection of bone marrow and blood samples at baseline, on days 30 and 100, and at 1 year. Patients undergo fluorothymidine F-18 PET, DECT, and water-fat MRI as in TMLI+FLT.

COHORT II (TBI): Patients undergo collection of bone marrow at baseline, day 30, time of relapse, and at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Cohort TMLI+FLT: AML patients eligible for and enrolling on COH 14012 or IRB 17505 that agree to participate in optional FLT PET imaging

  * Note: patients enrolling on IRB 19518 cannot enroll onto this cohort, but they may enroll on Cohort TMLI (below)
* Cohort TMLI: AML or ALL patients eligible for and enrolling on COH 14012, IRB 17505 or IRB 19518
* Cohort TBI: First or second remission AML or ALL patients that will receive TBI (13.2 Gy) plus chemotherapy (etoposide [VP16] 60 mg/kg or cyclophosphamide [Cy] 60 mg/kg for two days) as part of their standard of care
* Cohort TBI: Documented written informed consent of participant
* Cohort TBI: Age >= 18 to =< 60 years
* Cohort TBI: Patients who have not received a prior transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Change over time in cellularity and adiposity | Up to 1 year post-hematopoietic stem cell transplant (HCT)
  A non-parametric smoothing plot will be produced in the first step to view changes in the trend. Measurements will be summarized by mean +/- standard deviation (SD) at each time point. Exploratory within subjects' correlation will be examined using Pearson correlation between adjacent time points. A random-effects model will also be used to investigate whether there is significant time trend. Will use a two-sample t-test for comparing bone marrow cellularity percentage at pre-HCT and 1-year post-HCT between the total marrow and lymphoid irradiation (TMLI) group and total body irradiation (TBI) group (all cohorts). A paired t-test will also be carried out to examine if there is significant difference in changes of cellularity between these two groups.
Change over time of red marrow (cellularity) and yellow marrow (adipocyte) | Up to 2 years
  A non-parametric smoothing plot will be produced in the first step to view changes in the trend. Measurements will be summarized by mean +/- SD at each time point. Exploratory within subjects' correlation will be examined using Pearson correlation between adjacent time points. A random-effects model will also be used to investigate whether there is significant time trend. In addition, bone marrow/peripheral blood measurements will be correlated with survival outcome (relapse).
Number of hematopoietic stem cell (HSC) colony forming units (sub-analysis) | Up to 2 years
  Will be assessed by HSCs from marrow aspirate.
Ratio of HSC sub-populations (sub-analysis) | Up to 2 years
  Long-term, short-term, multi-potent progenitor, common myeloid progenitor, and granulocyte macrophage progenitor will all be assessed by HSCs marrow aspirate.
Hematopoietic stem cell density in bone marrow biopsy samples (sub-analysis) | Up to 2 years
  Will be assessed by CD34 staining.
Microvascular density in bone marrow biopsy samples (sub-analysis) | Up to 2 years
  Will be assessed by CD31 staining.

SECONDARY OUTCOMES:
Standardized uptake value (SUV) distribution at different skeletal sites | Baseline
  Changes in standardized uptake value (SUV) from fluorothymidine F-18 (FLT) positron emission tomography (PET) imaging uptake will be described. The distribution or heterogeneity will be first estimated using medians, ranges, interquartile ranges, means and standard deviations. Kolmogorov-Smirnov test (K-S) test will be performed to examine whether the distribution is the same for different skeletal sites. Also as a side product, sensitivity and specificity of the imaging will be estimated.
SUV distribution and presence of focal hot spot | Baseline
  Changes in SUV from FLT-PET imaging uptake will be described. The distribution or heterogeneity will be first estimated using medians, ranges, interquartile ranges, means and standard deviations. K-S test will be performed to examine whether the distribution is the same for different skeletal sites. Also as a side product, sensitivity and specificity of the imaging will be estimated.
Change in FLT PET activity | Baseline up to 2 years
SUVmax at site of biopsy | At time of biopsy
  SUVmax: the maximum SUV within the region of interest. SUVmin: the minimum SUV within the region of interest. SUVmean: the average SUV within the region of interest. As a primary goal we will be using SUVmax. Other parameters are secondary parameters.
  Sites: site of bone marrow biopsy is iliac crest. Image analysis is done at the different locations - iliac crest, Lumber spine, and femur.
SUVmean at site of biopsy | At time of biopsy
  SUVmax: the maximum SUV within the region of interest. SUVmin: the minimum SUV within the region of interest. SUVmean: the average SUV within the region of interest. As a primary goal we will be using SUVmax. Other parameters are secondary parameters.
  Sites: site of bone marrow biopsy is iliac crest. Image analysis is done at the different locations - iliac crest, Lumber spine, and femur.
Blast counts | Up to 2 years
  Will be assessed by bone marrow aspirate smears.
SUVmax at iliac crest, lumber spine, and femur | Up to 2 years
  For each location SUV measurement, software provides SUVmax, SUVmin and SUVmean. These are not separate measurements. Once region (volume) is defined, software will calculate SUV in the form of SUVmax, SUVmean and SUVmin. For simplicity, we will report SUVmax only as primary parameter. SUVmean and SUVmin will be secondary SUV parameters.
SUVmean at iliac crest, lumber spine, and femur | Up to 2 years
  For each location SUV measurement, software provides SUVmax, SUVmin and SUVmean. These are not separate measurements. Once region (volume) is defined, software will calculate SUV in the form of SUVmax, SUVmean and SUVmin. For simplicity, we will report SUVmax only as primary parameter. SUVmean and SUVmin will be secondary SUV parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States